CLINICAL TRIAL: NCT03088488
Title: Relationship of Bone Metabolism Biomarkers and Serum 25-Hydroxy Vitamin D in Patients With Chronic Periodontitis
Brief Title: Vitamin D and Periodontitis
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Cankat Kara, Professor, Ordu University
Other Study IDs: OrduUniversity
Record Dates: First submitted 2017-03-10; First posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Alveolar Bone Loss
Keywords: 25-OH vitamin D; RANKL; Osteoprotogerin; TNF-α
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Periodontally healthy subjects
  Interventions: Diagnostic Test: fasting venous blood samples
- Chronic periodontitis patients
  Interventions: Diagnostic Test: fasting venous blood samples

INTERVENTIONS:
Diagnostic Test: fasting venous blood samples

SUMMARY:
Vitamin D has become important for periodontal disease due to play a role in autoimmunity, bone mineral metabolism and inflammation. Our aim was to investigate the relation between serum 25-hydroxy vitamin D levels, clinical periodontal parameters and blood serum biomarkers. The subjects were evaluated in 2 groups as chronic periodontitis (n= 30) and periodontally healthy subjects (n= 30). Periodontal parameters and fasting venous blood samples were taken from the subjects to assess each patient's periodontal status and for biochemical analyses (25-hydroxy vitamin D (25-OH vit D), osteoprotegerin (OPG), receptor activator of nuclear kappa B ligand (RANKL), C-telopeptide (CTx), tumor necrosis factor-α (TNF-α)).

ELIGIBILITY:
* Inclusion Criteria:

  * never-smokers
  * no history of systemic disease
  * no patients had been under periodontal therapy and medicine for at least 6 months before the study
  * no pregnancy or lactation
  * no alcohol or antioxidant vitamin consumption.
* Exclusion Criteria:

  * -

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sixty patients (35 girls) who were aged between 25-45 years (30.8 (mean) ± 4.9 (standard deviation) and presented to our faculty for periodontal and other dental problems, participated in the study.
  Subjects were divided in to 2 groups each containing 30 patients:
  * Group I - periodontal healthy
  * Group II - untreated chronic periodontitis (radiographic evidence of bone loss and clinical attachment loss in excess of 5 mm in more than six teeth)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2016-04-21 (Actual)

PRIMARY OUTCOMES:
Biochemical parameters | Baseline
  serum TNF-α
Biochemical parameters | Baseline
  serum CTx
Biochemical parameters | Baseline
  serum RANKL
Biochemical parameters | Baseline
  serum OPG
Biochemical parameters | Baseline
  serum 25-OH vitamin D

SECONDARY OUTCOMES:
Periodontal parameters | Baseline
  The plaque index (PI)
Periodontal parameters | Baseline
  gingival index (GI)
Periodontal parameters | Baseline
  probing depth (PD)
Periodontal parameters | Baseline
  clinical attachment level (CAL)

IPD SHARING:
Plan to Share IPD: Undecided